CLINICAL TRIAL: NCT01967381
Title: Targeting GABA and Opioid Systems for a Pharmacotherapy for Methamphetamine Abuse
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Craig Rush, Professor, University of Kentucky
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R01DA033394 (NIH)
Record Dates: First submitted 2013-10-15; First posted 2013-10-22 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Methamphetamine Abuse; Methamphetamine Dependence
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Placebo Comparator): Subjects will be maintained on oral placebo.
  Interventions: Drug: Methamphetamine (Desoxyn®)
- Arm 2 (Experimental): Subjects will be maintained on oral oxazepam (Serax®).
  Interventions: Drug: Methamphetamine (Desoxyn®)
- Arm 3 (Experimental): Subjects will be maintained on oral naltrexone (Revia®).
  Interventions: Drug: Methamphetamine (Desoxyn®)
- Arm 4 (Experimental): Subjects will be maintained on oral naltrexone (Revia®) and oral oxazepam (Serax®).
  Interventions: Drug: Methamphetamine (Desoxyn®)

INTERVENTIONS:
Drug: Methamphetamine (Desoxyn®) — The pharmacodynamic effects of methamphetamine (Desoxyn®) will be determined during placebo, oxazepam (Serax®), naltrexone (Revia®) and combined oxazepam and naltrexone maintenance.

SUMMARY:
The research proposed in this application will determine the initial efficacy, safety and tolerability of a novel drug combination, oxazepam (Serax®) and naltrexone (Revia®), as a pharmacotherapy for methamphetamine (Desoxyn®) dependence. A rigorous, inpatient human laboratory study will be conducted. The proposed study is innovative and important because it will provide the impetus for the conduct of double blind, placebo-controlled trials to further demonstrate the efficacy of combined oxazepam and naltrexone for managing methamphetamine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime methamphetamine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to methamphetamine (Desoxyn®), oxazepam (Serax®) or naltrexone (Revia®)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Reinforcing Effects | After at least four days of placebo, oxazepam (Serax®), naltrexone (Revia®) or oxazepam and naltrexone maintenance
  The reinforcing effects of methamphetamine will be determined using a self-administration procedure in which subjects choose to take previously sampled doses. Reinforcing effects are measured during maintenance on placebo, oxazepam (Serax®), naltrexone (Revia®), and oxazepam and naltrexone combined.

SECONDARY OUTCOMES:
Subjective Effects | 12 sessions over approximately 4 week inpatient admissions
  Subjects will complete subjective effects measures during six sessions while they are admitted to our inpatient unit. These items will ask about drug effects and general mood.
Physiological and Side Effects | Daily over approximately 4 week inpatient admissions
  Physiological and side effects measures will be completed daily while subjects are admitted to our inpatient unit. Physiological measures include heart rate and blood pressure. Side Effects questions will query subjects about common effects of centrally active medications.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States